CLINICAL TRIAL: NCT05828680
Title: Circadian Rhythm Disruption in the Hospital Intensive Care Environment
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 852451
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective cardiac surgery
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
Abrupt changes to one's lifestyle disrupt biorhythms. Acute effects are well known from jet lag where transmeridian travel leads to insomnia, fatigue, irritability, gastrointestinal symptoms and other complaints. Several studies in the hospital environment reported dampened and misaligned biorhythms, suggesting that the inpatient experience is replete with circadian disruptors. However, comprehensive assessments of how circadian clocks are affected in intensive care and how this predicts post-operative recovery and risk are largely missing.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for cardiac surgery;
* ≥18 years of age;
* Capable of giving informed consent;
* Own a smartphone (Apple devices only).

Exclusion Criteria:

* Taking sleep aids (antihistamines, melatonin, etc.)
* History of alcohol abuse (more than 2 drinks a day with last drink within the past 3 days)
* History of substance abuse at risk of postoperative withdrawal;
* Active diagnosis of alcohol or substance abuse;
* Recent travel across more than two (2) time zones (within the past month);
* Planned travel across more than two (2) time zones during the planned study activities;
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
* Subjects without access to WiFi in their or close to home or at work;
* Patients with hearing aids;
* Heart transplant patients;
* Patients in isolation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential patients will be screened from outpatient clinic schedules from cardiac surgery appointments within the Perelman Center for Advanced Medicine. Patients for whom cardiac surgery is advised and who meet eligibility criteria will be approached and enrolled after their consultation with the surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sleep depth | Up to 48 hours
  Variance in sleep depth assessed as percent REM sleep of total sleep time (TST)

SECONDARY OUTCOMES:
Odds Ratio Product-based sleep depth | Up to 48 hours
  Variance in sleep depth assessed as Odds Ratio Product (ORP) which ranges between ORP=0 (deeply asleep) and ORB=2.5 (fully awake).
Cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | Up to 24 hours
  Variance in cognitive function
Number of recorded patient visits | 24 hours
  Any patient visits by physicians, nurses, maintenance and cleaning staff, family members and friends are documented
Purpose of recorded patient visits | 24 hours
  The rationale is documented descriptively for each patient visits by physicians, nurses, maintenance and cleaning staff, family members and friends

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skarke, MD, Principal Investigator — University of Pennsylvania; Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided